CLINICAL TRIAL: NCT00142467
Title: Phase II Study of Gemcitabine, Oxaliplatin in Combination With Bevacizumab (Avastin) in Patients With Hepatocellular Carcinoma
Brief Title: Gemcitabine, Oxaliplatin in Combination With Bevacizumab in Patients With Hepatocellular Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Dana-Farber Cancer Institute (Other); Beth Israel Deaconess Medical Center (Other); Brigham and Women's Hospital (Other); Genentech, Inc. (Industry); Sanofi-Synthelabo (Industry); Eli Lilly and Company (Industry)
Responsible Party: Principal Investigator, Andrew X. Zhu, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 03-390
Record Dates: First submitted 2005-08-31; First posted 2005-09-02 (Estimated); Last update posted 2014-03-18 (Estimated); Status verified 2014-03

CONDITIONS: Hepatocellular Carcinoma
Keywords: Unresectable hepatocellular carcinoma; Metastatic hepatocellular carcinoma; gemcitabine; oxaliplatin; bevacizumab; Avastin
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Gemcitabine; Oxaliplatin; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bevacizumab, Gemcitabine, Oxaliplatin (Experimental): For cycle 1 (14 days), bevacizumab 10 mg/kg was administered alone on day 1. For cycle 2 and beyond (28 days/cycle), bevacizumab 10 mg/kg was administered on days 1 and 15, gemcitabine 1,000 mg/m2 was administered as a dose rate infusion at 10 mg/m2/min followed by oxaliplatin at 85 mg/m2 on days 2 and 16. All drugs were administered intravenously until progression, intolerance, patient withdrawal, or death.
  Interventions: Drug: Gemcitabine; Drug: Oxaliplatin; Drug: Bevacizumab

INTERVENTIONS:
Drug: Gemcitabine
  Other Names: Gemzar
Drug: Oxaliplatin
  Other Names: Eloxatin
Drug: Bevacizumab
  Other Names: Avastin

SUMMARY:
The purpose of this study is to test the safety of bevacizumab when given in combination with gemcitabine and oxaliplatin and to see what effects (good or bad) it has on patients with hepatocellular carcinoma.

DETAILED DESCRIPTION:
* Treatment is given in cycles, each cycle (except for cycle 1) is 4 weeks long. Cycle 1 is only 2 weeks long.
* During cycle one only, bevacizumab will be given intravenously on day one. Two weeks after receiving bevacizumab, the patient will return to the clinic for treatment with all 3 study drugs.
* During cycle 2 and every cycle thereafter patients will receive; bevacizumab intravenously on day one and day 15; gemcitabine intravenously on day 2 and day 16; oxaliplatin intravenously on day 2 and day 16.
* The following evaluations will be conducted on day 1 and day 15 of each cycle (once every 2 weeks): physical examination, vital signs, medical history, blood tests and urine tests.
* Tumor measurements done by CT and/or MRI will be repeated at the end of cycle 3 and every 2 cycles thereafter.
* Dynamic Contrast-Enhanced Magnetic Resonance Imaging (DCE-MRI) of the liver and Perfusions CT scans will also be done on days 10-12 following bevacizumab treatment during cycle 1, and the Perfusion CT will be repeated at the end of cycle 3.
* Once study treatment is stopped the following evaluations will be performed: physical exam, vital signs, blood work, urine tests, CT scan of chest, abdomen and pelvis, and tumor measurements by CT or MRI scans.
* Follow-up will consist of physical examinations and blood tests every 6 months.
* Patients will continue to receive study treatment as long as there is no disease progression or unacceptable side affects.

ELIGIBILITY:
Inclusion Criteria:

* Unresectable or metastatic hepatocellular carcinoma
* Measurable tumors
* Adequate hepatic function: total bilirubin < 3.0mg/dl; AST < 7x ULN
* Adequate bone marrow function: ANC > 1,000/mm3; platelets > 75,000/mm3
* INR < 1.5 for those who are not on anticoagulation
* Up to two prior chemotherapy regimens for hepatocellular carcinoma
* 18 years of age or older
* ECOG performance status of 0-1
* Life expectancy of > 12 weeks

Exclusion Criteria:

* Clinically apparent central nervous system metastases or carcinomatous meningitis
* Uncontrolled serious medical or psychiatric illness
* Pregnant or lactating women
* Current or recent (within 4 weeks of first study infusion) participation in experimental study drug
* Uncontrolled hypertension
* Significant proteinuria
* Serious, non-healing wound, ulcer, or bone fracture
* Evidence of bleeding diathesis or coagulopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2004-04; Primary Completion 2006-08 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Time to disease progression of gemcitabine, oxaliplatin and bevacizumab regimen in patients with hepatocellular carcinoma. | 2 years
  From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years

SECONDARY OUTCOMES:
Number of participants with adverse events | 2 years
Objective response rate | 2 years
Overall survival | 2 years
  From date of randomization until the date of death from any cause, assessed up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Zhu, MD, Principal Investigator — Massachusetts General Hospital
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts